CLINICAL TRIAL: NCT00166114
Title: Do Antidepressants Reverse the Effects of Early Life Stress on the Brain and Thrombovascular System and Improve Psychological, Neuroendocrine, and Platelet Function: A Study of Men and Women With Childhood Abuse.
Brief Title: Depression, Epinephrine, and Platelet Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dominique Musselman, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0473-2002; 1R01HL065523-01A2 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Major Depressive Disorder
Keywords: platelet function; childhood abuse; depression; antidepressants; immune function; stress response
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Fractures, Stress | interventions — Escitalopram; Desipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram
- Desipramine (Active Comparator)
  Interventions: Drug: Desipramine

INTERVENTIONS:
Drug: Escitalopram — 10 mg of Escitalopram, and titrated up to 20 mg of Escitalopram after day 22 of intervention
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Desipramine — 25 mg of Desipramine for day 1-3, 50 mg of Desipramine for day 4-7, 75 mg of Desipramine for day 8-14, 100 mg of Desipramine for day 15-21. Titrated between 125 mg to 200 mg of Desipramine for day 22-56 of intervention
  Other Names: Norpramin
  Arms: Desipramine

SUMMARY:
Men and women who have suffered sexual and/or physical abuse before the age of 12 are at increased risk for anxiety and mood disorders, other serious psychiatric disorders, and likely medical illnesses. What is not known is whether adult survivors of childhood adversity experience heightened negative emotions and increased physical responses due to altered norepinephrine or serotonin systems in their brains and bodies. The investigators expect to see that survivors of childhood adversity experience heightened negative emotions and increased physical responses to stress.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Individuals who are suicidal, psychotic, or with bipolar depression
* alcohol or substance abuse or
* regularly use medications which alter mood or blood vessel function (zolpidem or zalpelon, aspirin, nonsteroidal antiinflammatory drugs, sympatholytics, theophylline, central acting agonists, beta-blockers, coumadin, nitrates, triazolobenzodiazapines, or use steroids (testosterone-patch or pill form), use tryptophan or monoamine oxidase inhibitors (MAOIs),
* have narrow-angle glaucoma, liver disease,
* severe allergies (especially to antidepressants similar to escitalopram or desipramine)
* seizures, or a serious medical disorder (e.g. hypothyroidism) that is unstable or is untreated.
* Depressed patients with a prior history of severe adverse events associated with SSRIs or TCAs will not be accepted into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L Musselman, MD,MS, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Background] Royster EB, Trimble LM, Cotsonis G, Schmotzer B, Manatunga A, Rushing NN, Pagnoni G, Auyeung SF, Brown AR, Schoenbeck J, Murthy S, McDonald WM, Musselman DL. Changes in heart rate variability of depressed patients after electroconvulsive therapy. Cardiovasc Psychiatry Neurol. 2012;2012:794043. doi: 10.1155/2012/794043. Epub 2012 Aug 27. PMID 22966422
- [Background] Shively CA, Musselman DL, Willard SL. Stress, depression, and coronary artery disease: modeling comorbidity in female primates. Neurosci Biobehav Rev. 2009 Feb;33(2):133-44. doi: 10.1016/j.neubiorev.2008.06.006. Epub 2008 Jun 24. PMID 18619999
- [Background] Bruce EC, Musselman DL. Depression, alterations in platelet function, and ischemic heart disease. Psychosom Med. 2005 May-Jun;67 Suppl 1:S34-6. doi: 10.1097/01.psy.0000164227.63647.d9. PMID 15953798
- [Result] Bruce EC, Guo Y, Lawson KC, Manatunga AK, Auyeung SF, McDonald WM, Rushing N, Brown AR, Gilles N, Emery M, Bonsall R, Porquez J, Stowe Z, Nemeroff CB, Musselman DL. Platelet thromboxane A2 secretion in patients with major depression responsive to electroconvulsive therapy. Psychosom Med. 2008 Apr;70(3):319-27. doi: 10.1097/PSY.0b013e3181663580. Epub 2008 Mar 31. PMID 18378867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from Emory Psychiatry Clinic outpatient population
Groups:
- Escitalopram: Subjects received 10 mg of Escitalopram for 22 days and then were titrated up to 20 mg of Escitalopram after day 22 of intervention until day 56
- Desipramine: Subjects received 25 mg of desipramine for day 1-3, 50 mg of desipramine for day 4-7, 75 mg of desipramine for day 8-14, 100 mg of desipramine for day 15-21. Subjects titrated between 125 mg to 200 mg of desipramine for day 22-56 of intervention
Period: Overall Study
Arm/Group | Escitalopram | Desipramine
Started | 21 | 19
Completed | 7 | 13
Not Completed | 14 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Escitalopram: Subjects received 10 mg of Escitalopram for 22 days and then were titrated up to 20 mg of Escitalopram after day 22 until day 56
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Desipramine | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants] — Age, Categorical
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 21 | 19 | 40
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Response of Participants, Defined by Change in the 21-item Hamilton Depression Rating Scale (HDRS) From Baseline to Week8
Description: Number of subjects that showed no response, partial response, and response based on scores from baseline and week 8.
  The 21-item HDRS measures depression severity. The scoring is sum the total of all 21 items to arrive at the total score, with a range of 0 to 60, where higher scores indicated greater severity. Nine items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Eleven items are scored from 0 - 2 (0 = absent and 2 = severe). The last item is scored on a 4-point scale of 0-3 (0 = absent and 3 = severe). The HDRS at week 8 was compared to the baseline HDRS and each participant's response was calculated using the below table:
  No Response = < 25% change in Depression Rating Scale Score Partial Responder = < 50% to >25% change in Depression Rating Scale Score Responder = 50% or greater change in Depression Rating Scale Score
Time Frame: Baseline, Week 8
Measure: Number; unit: participants
Arm/Group | Escitalopram | Desipramine
Number analyzed (Participants) | 7 | 13
participants
  Response | 5 | 9
  No or Partial Response | 2 | 4
Statistical Analysis 1: Comparison: Escitalopram; Chi Square test was performed comparing actual vs. expected non- and partial response or response to either escitalopram or desipramine treatment; Test type: Superiority or Other; p = .918, Chi-squared

ADVERSE EVENTS:
Arm/Group | Escitalopram | Desipramine
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/19
Other Adverse Events (participants affected / at risk) | 13/21 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=21) | Desipramine (N=19)
Suicide gesture (superficial lacerations to wrists with a razor) (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=21) | Desipramine (N=19)
Dry Mouth (Skin and subcutaneous tissue disorders) | 2 | 2
Orthostatic Tachycardia (Cardiac disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Stomach Pain (Gastrointestinal disorders) | 0 | 1
Indigestion (Gastrointestinal disorders) | 1 | 1
Increased Liver Function Test (Metabolism and nutrition disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 1 | 1
Sedation (Nervous system disorders) | 1 | 0
Fatigue (Nervous system disorders) | 2 | 0
Insomnia (Nervous system disorders) | 0 | 1
Weight Loss (Metabolism and nutrition disorders) | 0 | 1
Confusion (Nervous system disorders) | 1 | 0
Irritability (Nervous system disorders) | 1 | 0
Ejaculation Disorder (Reproductive system and breast disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No